CLINICAL TRIAL: NCT00352391
Title: Vanguard Study Characterizing Occurrence of Recurrent or Second Primary Tumors in Patients With Prior History of Definitively Treated Stage I/II Head and Neck or Non-Small Cell Lung Cancer Who Are Current or Former Smokers
Brief Title: Vanguard Study for Head and Neck Cancer or Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2003-0424
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Head And Neck Cancer; Lung Cancer; Bronchoscopy; Laryngoscopy; NSCLC; Disease Free Survival; Current Smoker; Former Smoker
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of lung tissue, saliva, blood, and scrapings from inside of cheek. Fluid and mucous collected during bronchoscopies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vanguard Study: Patients with Head and Neck or Non-Small Cell Lung Cancer who are Current or Former Smokers.
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — At Months 6, 12, 18, 24, 30, and 36, complete medical history will be recorded, and a physical exam will be performed by either a doctor or a nurse. At each of these visits, blood will be drawn for routine tests (about 3 teaspoons) and for research purposes (about 4 teaspoons). Also, a chest x-ray and a chest CT will be done at these visits.

SUMMARY:
The goal of this research study is to look at how long individuals who have been treated for early stage NSCLC or HNSCC live without developing lung cancer. Another goal is to develop tools to help predict the likelihood of lung cancer occurrence in this population. This will be done by studying characteristics of tissue and bodily fluids (including blood).

Objectives:

* To assess the smoking-related disease-free survival in patients who are current or former smokers with a prior definitively-treated stage I/II lung or head and neck cancer.
* To develop a risk model to help predict the likelihood of lung cancer development both imaging and biomarker based in this high-risk population.

DETAILED DESCRIPTION:
This study is known as the Vanguard Trial. When you enter this study, you will have a complete medical history (including smoking history) and physical exam, including measurement of height, weight, and vital signs (including blood pressure, heart rate, and temperature). You will have a performance status evaluation (a test looking at the ability to perform every day activities). You will have blood samples drawn for routine blood tests (about 3 teaspoons), to check your blood clotting function (about 1-2 teaspoons), and for research purposes (about 4 teaspoons). You will have a chest x-ray and a CT scan of your chest. Women who are able to have children must have a negative blood or urine pregnancy test. If you are currently a smoker, you will be given information on programs to help you quit smoking. Although you will be encouraged to quit smoking, you do not have to quit smoking or participate in these programs to be a part of this study.

You will also have a bronchoscopy (tissue sample from the lung) at the beginning of this study for lab analysis. For this procedure, you will be given drugs to relax. Then, a local anesthetic will be sprayed in your nose and throat to numb those areas. A slim, flexible tube with a light will be placed through your nose or mouth and into your lungs. Tweezers will be fed through the tube to collect lung tissue (biopsy) samples from 6 different places in your lungs. During the bronchoscopy procedure, a complete inspection of the airways will be performed. Any suspicious areas that are seen under the white-light and autofluorescence bronchoscopy will be identified and more biopsies and brushings will be performed to evaluate whether any pre-cancerous tissue is present. You will also have a bronchial brushing next to each biopsy site. In a bronchial brushing, a small brush is fed through the tube into your lungs and a sample of lung tissue is gently scraped off. When the biopsies and brushings are done, you will have a bronchial lavage (bronchial washing). In the bronchial lavage, a small amount of water (about 4 tablespoons) is sprayed into your lungs and then suctioned out through the tube. This fluid is used to collect additional tissue and mucous samples. In addition, a sputum (saliva) sample will be taken and the inside of your cheek will be scraped (buccal sample).

If you have had HNSCC, you will also have a laryngoscopy. In a laryngoscopy, a lighted tube is placed down your throat and the larynx is checked. The back of your throat will be sprayed with an anesthetic before this procedure to make the procedure more comfortable.

While on study, you will return to the clinic for at least 3 years and for up to a total of 6 years. At Months 6, 12, 18, 24, 30, and 36, your complete medical history will be recorded, and you will have a physical exam by either a doctor or a nurse. At each of these visits, you will also have blood drawn for routine tests (about 3 teaspoons) and for research purposes (about 4 teaspoons). You will also have a chest x-ray and a chest CT at these visits. At Months 12, 24 and 36, you will have blood drawn (about 1-2 teaspoons) to check your blood-clotting function. If you think you may be pregnant, you will also have a urine or blood pregnancy test. In addition, you will have a bronchoscopy and provide sputum and buccal smear samples at your 12 month visit. If you have been treated for HNSCC you will have a laryngoscopy at 12 months.

You have the right to leave the study at any time. If you choose to stop participating in this study, you will be asked to return to the clinic for a final clinic visit. At this visit, your complete medical history will be recorded, and you will have a physical exam and blood drawn for routine tests (about 3 teaspoons) and for research purposes (about 4 teaspoons). Your study doctor will also ask you about your current smoking use, any medications you are taking, and how you are feeling (symptoms).

This research study includes two bronchoscopies done one year apart. These bronchoscopies are being done primarily for research purposes and are unlikely to provide information useful in your individual treatment. These bronchoscopies do have risks associated with them. These risks are described in section 4 of this informed consent document.

Recent research on early stage NSCLC indicates that adjuvant chemotherapy after surgery increases the length of time a person may survive and the length of time before cancer recurs. However, this adjuvant chemotherapy also has side effects that can be severe and in rare cases fatal. If you have had surgery for NSCLC and wish to receive adjuvant chemotherapy, you may only enroll in the Vanguard study after you have completed the adjuvant chemotherapy.

As part of this study you will provide samples of your lung tissue, saliva, blood, and scrapings from the inside of your cheek. Fluid and mucous collected during the bronchoscopies will also collected. These samples will be studied by scientists to learn about genes and proteins in people who have been treated for early NSCLC or HNSCC. The samples will also be used to grow cells and cultures that will be used to test chemotherapy drugs. These cells and cultures will also be used to learn about genes and proteins.

All M. D. Anderson researchers are trained in the importance of maintaining patient privacy. Your privacy will be protected by assigning you a number that will be used in place of your name on documents that are part of this study. A list that links your name with your study number will be stored in a restricted file that may be accessed only with a password. Only a few essential research personnel have access to this password.

At the end of the study you will not be automatically notified of the research findings. If you wish to learn about the results, however, you may request them from the principal investigator:

Principal Investigator: Waun Ki Hong, MD 1515 Holcombe Blvd., Unit 432 MD Anderson Cancer Center Houston, TX 77030

This is an investigational study. A total of about 50 individuals will take part in this study. Participants will be enrolled at M. D. Anderson and several other sites around the country.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either: a) histologically proven stage I, II, IIIa NSCLC who have undergone a complete surgical resection of the primary tumor OR b) stage I or II HNSCC who have undergone definitive local treatment (surgery or radiation therapy).
2. HNSCC patients:Definitive local treatment </= 12 months prior to trial enrollment. NSCLC patients: Surgery </= 12 months prior to trial enrollment.
3. No evidence residual cancer
4. Age > = 18 years
5. Performance status of 0- 2 (Zubrod)
6. Patients must have no contraindications for undergoing bronchoscopy.
7. Patients must have no active pulmonary infections.
8. Participants must have the following blood levels: total granulocyte count >1500; platelet count > 100,000; total bilirubin < = 1.5 mg. %; and creatinine < = 1.5 mg %.
9. Participants must complete the pretreatment evaluation and must consent to bronchoscopy and to endobronchial biopsy for biomarker studies.
10. All subjects who agree to participate will be given a written and verbal explanation of the study requirements and a consent form that must be signed prior to registration. Subjects will be informed that (a) they must be willing to take biopsies through bronchoscopy and give blood samples at the specified times, (b) they must schedule and keep the specified follow-up visits with their physicians and the study clinics, and (c) side effects and health risks may occur, as described in the informed consent form.
11. Smoking history of at least 10 pack years. May be current or former smoker.
12. Subject must be considered legally capable of providing his or her own consent for participation in this study.
13. HNSCC patients only: Must have no contraindications for undergoing laryngoscopy.

Exclusion Criteria:

1. History of radiation therapy to the chest. For those patients with head and neck cancer who received radiation, no more than 10% of the lung volume (apices) may be included.
2. History of systemic chemotherapy. Exception: NSCLC patients may have had up to 4 cycles of platinum-based doublet therapy.
3. Pregnant or breast-feeding (a negative pregnancy test within 72 hours of enrollment for women with child-bearing potential is required).
4. Participants with active pulmonary infections or recent history of pulmonary infection (within one month).
5. Participants with acute intercurrent illness.
6. Participants requiring chronic ongoing treatment with NSAIDs except aspirin.
7. Participants with history of stroke, uncontrolled hypertension, and/or uncontrolled angina pectoris.
8. Patients may not take high dose antioxidants (vitamins E or C) during the study period. "High dose" will be determined by the study investigators.
9. Patients may not take high dose synthetic or natural Vitamin A derivatives (> 10,000 IU per day). "High dose" is defined as anything greater than a once-daily multivitamin. Any additional supplementation will be evaluated at the discretion of the treating physician.
10. History of biologic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a prior history of a definitively treated stage I/II head and neck or non-small cell lung cancer who are current or former smokers.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2004-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Smoking-Related Disease-Free Survival (S-DFS) | 6 Years
  Smoking-related disease-free survival (S-DFS) defined as time from registration to the development of recurrence, smoking related SPT, or disease-specific death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: George Simon, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Conemaugh Memorial Medical Center, Johnstown, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org